CLINICAL TRIAL: NCT02571699
Title: Minimum Effective Volume of Lidocaine-Bupivacaine for Ultrasound-Guided Subgluteal Sciatic Nerve Block
Brief Title: Minimum Effective Volume of Lidocaine-Bupivacaine for Subgluteal Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, De Tran, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGH
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Injuries to the Ankle and Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subgluteal sciatic block (Active Comparator): Subgluteal block with similar volume
  Interventions: Other: Subgluteal Nerve Block
- Subgluteal block (Experimental): Subgluteal block with decreasing volume
  Interventions: Other: Subgluteal Nerve Block

INTERVENTIONS:
Other: Subgluteal Nerve Block — ultrasound-guided subgluteal sciatic nerve block.

SUMMARY:
The aim of this study is to determine the minimum effective volume of LA in 90 % of patients (MEV90) required for US-guided subgluteal sciatic nerve block.

DETAILED DESCRIPTION:
The aim of this study is to determine the minimum effective volume of LA in 90 % of patients (MEV90) required for US-guided subgluteal sciatic nerve block.

Success rate is defined as a minimal composite score of 6 points (out of 8 points) at 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 35

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets≤ 100, International Normalized Ratio≥ 1.4 or partial prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to LA
* pregnancy
* prior surgery in the subgluteal region
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
success rate | 0-30 minutes
  minimal composite score of 6 out of 8 points

CONTACTS AND LOCATIONS:
Overall Officials: De Tran, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada